CLINICAL TRIAL: NCT07325266
Title: Human Laboratory Study of Apremilast for Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HLAB-004
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Alcohol Misuse
MeSH Terms: conditions — Alcoholism | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Apremilast 60 mg/day (Active Comparator): Apremilast, 30mg per capsule, administered twice daily (AM/PM), Placebo, administered once daily (AM)
  Interventions: Drug: Apremilast
- Oral Apremilast 90 mg/day (Active Comparator): Apremilast, 30mg per capsule, 2 capsules (AM) and 1 capsule (PM)
  Interventions: Drug: Apremilast
- Oral Matched Placebo (Placebo Comparator): Placebo, capsule, 2 capsules (AM) and 1 capsule (PM)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matched Placebo Capsule
  Arms: Oral Matched Placebo
Drug: Apremilast — 30 mg capsule
  Other Names: Otezla
  Arms: Oral Apremilast 60 mg/day; Oral Apremilast 90 mg/day

SUMMARY:
Primary: The primary objective of this study is to compare the efficacy of two different maintenance doses of apremilast (tablets) in reducing alcohol craving among subjects with moderate to severe alcohol use disorder (AUD) after two weeks of daily dosing.

Secondary: Secondary objectives include evaluation of two different maintenance doses of apremilast compared with matched placebo on other measures of self-reported alcohol consumption, alcohol craving, alcohol-related negative consequences, AUD symptoms, pain, sleep disturbances, depression, anxiety, quality of life, cigarette smoking, other nicotine use, cannabis use, retention in the study, and safety.

ELIGIBILITY:
Inclusion Criteria (not exhaustive list):

1. Be at least 21 years of age.
2. Have a current (past 12 months) DSM-5 diagnosis of AUD (4 or more symptoms) assessed using the MINI neuropsychiatric interview version 7.0.2 (at least moderate severity).
3. Have a BAC by breathalyzer equal to 0.000 when s/he signed the informed consent document (either just prior to or immediately after signing consent).
4. Be seeking treatment for problems with alcohol and express a goal of abstinence or a reduction in drinking.
5. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
6. Agree (if the participant is female and of childbearing potential) to use at least one of the following methods of birth control, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal:

   * oral contraceptives,
   * contraceptive sponge,
   * patch,
   * double barrier (diaphragm/spermicidal or condom/spermicidal),
   * intrauterine contraceptive system,
   * etonogestrel implant,
   * medroxyprogesterone acetate contraceptive injection,
   * complete abstinence from sexual intercourse, and/or
   * hormonal vaginal contraceptive ring.
7. Be willing to adhere to the investigational product dosing schedule.
8. Complete all assessments required at screening and baseline.
9. Have a place to live in the 2 weeks prior to randomization and not be at risk that s/he will lose his/her housing by Study Week 6.
10. Not anticipate any significant problems with transportation arrangements or available time to travel to the study site by Study Week 6.
11. Not have any plans to move within Study Week 6 to a location which would make continued participation in the study impractical.
12. Provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the participant in case of a missed clinic appointment.
13. Be someone who in the opinion of the investigator would be expected to complete the study protocol.
14. Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may substantially interfere with study participation.
15. If taking a medication for depression, must have been taking a stable dose in the 2-months prior to randomization and plan to continue during the study. This includes drugs such as the following:

    * SSRIs
    * Dual uptake inhibitors
    * SNRIs
    * Tricyclic antidepressants
    * MAOIs
    * Bupropion
16. Not currently taking apremilast and agree not to take non-study supplied apremilast for the duration of the study.
17. Have normal renal function defined as creatinine clearance ≥ 60 mL per minute by the Cockcroft-Gault equation.

Exclusion Criteria:

Contact study site for exclusion criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol Craving | Week 4
  The primary outcome measure of this study is to compare the efficacy of two different maintenance doses of apremilast (tablets) in reducing alcohol craving among participants with moderate to severe alcohol use disorder (AUD) after two weeks of daily dosing.

SECONDARY OUTCOMES:
Participants with no heavy drinking days | Weeks 2-5
  Percentage of participants with no heavy drinking days over the last 4 weeks of the treatment period. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
Participants abstinent from alcohol | Weeks 2-5
  Percentage of participants abstinent from alcohol over the last 4 weeks of the treatment period of treatment.
Days abstinent from alcohol per week. | Weeks 2-5
  Percentage of days abstinent from alcohol per week.
Participants with at least a WHO 2-level decrease in alcohol consumption | Weeks 2-5
  Percentage of participants with at least a WHO 2-level decrease in alcohol consumption
Heavy drinking days per week | Weeks 2-5
  Percentage of heavy drinking days per week
Participants abstinent from cigarette smoking | Weeks 4-5
  Percentage of participants abstinent from cigarette smoking (among smokers at baseline)
Number of drinks per week | Weeks 2-5
  Mean number of drinks per consumed week
Number of drinks per drinking day | Weeks 2-5
  Weekly mean number of drinks consumed per drinking day.
Alcohol Use Disorder Symptoms | Week 6
  Number of Alcohol User Disorder (AUD) symptoms as measured by MINI AUD
Number of days of cannabis use per week | Weeks 4-6
  Mean number of days of cannabis use per week (among cannabis users at baseline)
Global Health Score | Weeks 4,6
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health Scale is QOL assessment to evaluate the clinical benefit of apremilast treatment. It is a 10-question self-report measure that rates items on a 5-item ordinal scale (5 = Excellent, 1 = Poor) over the past 7 days. It assesses five core health domains: physical function, pain, fatigue, emotional distress, and social health. Scores will be converted to T-scores (normalized for comparison across populations). Lower scores correspond to more severe problems. Global health score measured by the PROMIS-Global Health scale
Alcohol Negative Consequences Score | Weeks 4,6
  For negative consequences for alcohol use, the short form of the PROMIS Patient-Reported Outcomes Measurement Information System) Alcohol Negative Consequences questionnaire will be used to assess outcomes of alcohol use over the past 7 days. This 7-item questionnaire assesses physical and social consequences of drinking. Scores will be converted to T-scores (normalized for comparison across populations).
Sleep Disturbance | Weeks 4,6
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbances Scale - short form is an 8-item scale asking questions about sleep disturbances in the past 7-days. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance. Scores will be converted to T-scores (normalized for comparison across populations).
PROMIS pain intensity score | Weeks 4,6
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Adult Short Form version 1.0 Pain Intensity will be used to assess pain intensity using a 7-day recall period (2 items) and pain intensity right now (1 item). Each item has a 5-point scale with anchors at "had no pain" and "very severe". The responses to each item will be summed to calculate a total pain intensity score. Scores will be converted to T-scores (normalized for comparison across populations).
PROMIS-Anxiety Scale score | Weeks 4-6
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety Scale - short form is a 8-item scale asking questions about anxiety in the past 7 days with anchors at 1 (never) and 5 (always). Interpretation of scoring is as follows:
  Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
  Scores will be converted to T-scores (normalized for comparison across populations).
HAM-D17 score | Weeks 2,4,6
  A 17-item clinician administered Hamilton Depression scale (HAM-D17) will be used to monitor the development of depressive symptom throughout the study. A structed interview guide must be followed by the administrator performing this assessment.
  HAM-D17 scores of below 7 (no depression), 7 to 17 (mild depression), 18 to 24 (moderate depression) and 25 and above (severe depression) (Carrozzino-2020). This questionnaire will be completed by the interviewer and will be both the source and eCRF.
Urge to Drink scale scores | Weeks 2-5
  Urge to Drink craving score during the minimum period. Minimum score of = 0 and maximum = 35
Inflammatory Markers | Weeks 3, 6
  Clinical chemistry and hematology laboratory tests will be performed at the clinical site's local clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Falk, PhD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (3):
- United States (3):
  - University of California, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Virginia, Charlottesville, Virginia